CLINICAL TRIAL: NCT07055477
Title: A Phase I Trial of Anti-CC Chemokine Receptor 4 Chimeric Antigen Receptor T Cells (CCR4 CAR T Cells) for CCR4 Expressing T-cell Malignancies Including Peripheral T-cell Non-Hodgkin Lymphoma (PTCL) and Cutaneous T-cell Non-Hodgkin Lymphoma (CTCL)
Brief Title: A Phase I Trial Anti-CC Chemokine Receptor 4 Chimeric Antigen Receptor T Cells (CCR4 CAR T Cells) for CCR4 Expressing T-cell Malignancies Including Peripheral T-cell Non-Hodgkin Lymphoma (PTCL) and Cutaneous T-cell Non-Hodgkin Lymphoma (CTCL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001774; 001774-C
Record Dates: First submitted 2025-07-08; First posted 2025-07-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Relapsed and/or Refractory Mature T Cell Malignancy; Peripheral T-Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Hepatosplenic T-cell Lymphoma; Monomorphic Epithelialtropic Intestinal Lymphoma; Enteropathy Associated T-cell Lymphoma; Cutaneous T-Cell Lymphoma; Mycosis Fungoides; Subacute Panniculitis-like T-cell Lymphoma
Keywords: CCR4; CAR T; Chemokine Receptor 4; Chimeric Antigen Receptor; Gene Therapy; Cell Therapy; Immunotherapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Conditioning chemotherapy with cyclophosphamide and fludarabine followed by autologous CCR4 CAR T-cells (IV) at escalating doses
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Autologous CCR4 CAR T cells
- Arm 2 (Experimental): Conditioning chemotherapy with cyclophosphamide and fludarabine followed by autologous CCR4 CAR T-cells (IV) at the MTD
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Autologous CCR4 CAR T cells

INTERVENTIONS:
Drug: Cyclophosphamide — Days -5 to -3: Cyclophosphamide 300 mg/m^2 x 3 days
Drug: Fludarabine — Days -5 to -3: Fludarabine 30 mg/m^2 IV daily over 30 minutes for 3 days
Biological: Autologous CCR4 CAR T cells — Day 0: Cells will be infused intravenously (IV) over 10-30 minutes

SUMMARY:
Background:

Chemokine receptor 4 (CCR4) is a protein that is found on the surface of certain T-cell lymphoma cells and is common in mature T-cell cancers. White blood cells can be changed with molecules called anti-CCR4 to express a chimeric antigen receptors (CAR), which is a molecule that directs a white blood cell to attack other cells. The CAR in this study attacks the CCR4 protein found on your T-cell lymphoma. This type if therapy is called gene therapy. Gene therapy involves a person s own white blood cells modified to target cancer cells. More research is needed to find out if gene therapy can treat T-cell cancers and do it safely.

Objective:

To test safety of giving people with certain mature T-cell lymphomas their own white blood cells modified with anti-CCR-4 CAR.

Eligibility:

People aged 18 and older with certain mature T-cell lymphomas that have not responded to or have come back after treatment. They must have a T-cell lymphoma that has CCR4 on the surface of the cancer cells.

Design:

Participants will be screened. They will have a medical history and physical exam. Tests of blood, urine, and heart and lung function will be done.

Participants will have tests:

Computed tomography (CT), positron emission tomography (PET), and magnetic resonance imaging scans: They will lie on a table that slides into a donut-shaped machine or a tube. Pictures of the inside of the body will be taken. Before the PET scan, they will get an injection of radioactive fluid in a vein in the arm. Before the MRI, they may get a contrast dye injected through a vein (IV) in the arm.

A biopsy of the tumor may be taken. A bone marrow sample may be taken from the hip: The area will be numbed and a large needle inserted through the skin.

Leukapheresis will be done to obtain T-cells that will be genetically modified to express anti-CCR4 CARs on T-cells: Blood is drawn through an IV in one arm, circulated through a machine, and then returned through an IV in the other arm.

Chemotherapy drugs will be given in an IV to prepare the body to accept the modified CAR T cells.

The modified cells will be given in an IV.

Participants will be followed for 15 years: This will require blood tests over the first 1-2 years followed by yearly visits and possibly telehealth updates....

DETAILED DESCRIPTION:
Background:

* Chemokine receptor 4 (CCR4) the receptor for C-C chemokines CCL17 [Thymus and activation-regulated chemokine (TARC)] and CCL22 [Macrophage-derived chemokine (MDC)] is expressed on some subsets of normal human T lymphocytes including T regulatory cells (Tregs), TH2 and TH17 cells. It is also widely expressed in mature T-cell malignancies.
* The anti-CCR4 antibody, mogamulizumab, has shown appreciable clinical activity against CCR4 expressing T-cell malignancies suggesting this molecule to be a robust therapeutic target.
* A lentivirus vector-based 2nd generation anti-CCR4 chimeric antigen receptor (CCR4-CAR.4-1BB-CD3Zeta) has been generated, and its functionality and specificity have been validated in in-vitro cell lysis assays with several patient-derived CCR4+ malignant T cells lines as has its efficacy in a murine xenograft preclinical model of ATL.

Objectives:

-Determine safety of administering autologous CCR4 CAR T cells.

Eligibility:

* Diagnosis of relapsed/refractory mature T cell malignancy that expresses CCR4 including: Peripheral T-cell Lymphoma not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL), hepatosplenic T-cell lymphoma (HSTCL), monomorphic epithelialtropic intestinal lymphoma (MEITL), enteropathy associated T-cell lymphoma (EATL) or cutaneous Tcell lymphoma (CTCL) including mycosis fungoides and subacute panniculitis-like Tcell Lymphoma or lymphomatous subtypes of ATL without evidence of CNS involvement or substantial circulating disease.
* Age >=18 years.
* Adequate organ function and absence of medical conditions that would preclude safe administration of this treatment.

Design:

* Single-institution, open-label, non-randomized, 3+3 pilot dose escalation trial
* Participants will undergo leukapheresis to obtain T-cells that will be genetically modified to express anti-CCR4 CARs on T-cells. Groups of 3 to 6 participants will receive autologous CCR4 CAR T cells at doses of 0.3 x 10^6/kg, 1 x 10^6/kg and 3 x 10^6/kg provided that DLT has not been reached; If the first dose level exceeds the MTD, a subsequent cohort of 3-6 participants will be treated at the dose level of 0.1 x 10^6/kg.
* Up to 9 additional participants will be treated at the MTD or the maximum administered dose to better assess the activity of this treatment regimen.
* Participants will be monitored for toxicity, antitumor effects and persistence of CCR4 CAR T-cells and assessed for response with periodic re-staging imaging and laboratory testing.
* Statistical analyses will be limited to summary statistics by dose level and for all participants for safety parameters, biologic effects, response rate and survival.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Pathologically (biopsy) confirmed histologic diagnosis of a relapsed/refractory CCR4+ mature T-cell malignancy from one of the following subtypes: peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL), hepatosplenic t-cell lymphoma (HSTCL), monomorphic epithelialtropic intestinal lymphoma (MEITL), enteropathy associated T-cell lymphoma (EATL) or cutaneous T-cell lymphoma (CTCL) including mycosis fungoides and subacute panniculitis-like T-cell Lymphoma, or lymphomatous subtypes of ATL without evidence of CNS involvement or substantial circulating disease confirmed by the Laboratory of Pathology, NCI.

  --CCR4+ is defined as >= 10% malignant cells positive for CCR4 by immunohistochemistry. It is preferred to have a fresh biopsy to confirm the CCR4 status. In the event a fresh biopsy cannot be safely performed in the opinion of the treating physician, an archival biopsy sample taken at the time of previous progression can be used.
* Adequate tissue [a formalin fixed tissue block or 15 slides of tumor sample (archival or fresh)] from diagnostic biopsy (archival or fresh) must be available.

NOTE: Tissue will be used for assessment of CCR4 expression on malignant cells by immunohistochemistry with any leftover slides or samples to be used for correlative studies. Tumor tissue may be from any previously collected tissue and adequacy is at the discretion of the Principal Investigator. If prior tissue is not available, a screening biopsy will be necessary unless repeat biopsy is deemed unsafe by the treating physician in consultation with the Principal Investigator.

* Participants must have disease that is relapsed or refractory after prior therapy as follows:

  * Participants with ALCL must have failed at least one prior line of Brentuximab-containing therapy.
  * Due to the generally indolent nature of the disease, participants with Mycosis Fungoides must have exhausted all standard therapies as determined by the enrolling physician and principal investigator to be eligible for this study.
  * All other participants must have failed at least two lines of prior therapy.
* Participants must have measurable or evaluable disease at the time of enrollment. For participants with systemic T-cell lymphoma, this is defined by any evidence from CT scan or PET-CT-avid disease based on the Lugano criteria. For participants with Cutaneous T-cell Lymphoma, positive scores based on Modified Severity-Weighted Assessment Tool (mSWAT) criteria are acceptable.
* Participants must be >=18 years of age at the time of signing informed consent.
* Adequate performance status (PS) as follows: ECOG PS 0-1.
* Adequate organ function as evidenced by the following laboratory parameters:

  * Absolute neutrophil count (ANC) >= 1,000 /microL
  * Platelets >= 75,000 / microL
  * Hemoglobin (Hgb) >= 9 g/dL (transfusions permitted)
  * Creatinine Clearance >= 60 mL/min/1.73m^2 per Cockcroft Gault equation; For participants < 60 per Cockcroft Gault a direct measurement may be used
  * Serum total bilirubin <= 3 X upper limit of normal (ULN)
  * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) <= 3 X ULN
  * Left ventricular ejection fraction > 50% by echocardiogram performed
  * ECG No clinically significant ECG findings (Arrhythmias or evidence of ischemic heart disease with clinical correlate)

Note: Participants with well-controlled atrial fibrillation are eligible.

--FEV1 and DLCO > 60% of predicted (adjustment for Hgb acceptable)

-Individuals of child-bearing potential (IOCBP) must have a negative urine or blood HCG pregnancy test at screening.

NOTE: IOCBP is defined as any person assigned female at birth who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

-Individuals of child-bearing potential (IOCBP) must agree to use highly effective contraception (hormonal, intrauterine device [IUD], abstinence, surgical sterilization) or practice abstinence starting at the time of study entry, for the duration of study therapy, and 12 months after the last dose of combined chemotherapy.

Individuals able to father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and for 4 months after the last dose of combined chemotherapy. We also will recommend these individuals with partners of childbearing potential ask partners to be on highly effective birth control (hormonal, IUD, surgical sterilization)

* Nursing participants must be willing to discontinue nursing through 12 weeks after cell infusion.
* Potential participants must agree to stay within 1-hour drive of NIH clinical center from date of initial discharge from hospitalization (no earlier than D+15) through initial D+28 follow-up and be willing and able to return for in-person follow-up visits through month 3 of the study.
* Ability of participant or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with any current or prior CNS involvement by malignancy are excluded from this study. All potential participants will be screened with brain imaging prior to enrollment on study.
* Participants with >1000 atypical cells/mm^3 by peripheral blood flow cytometry at screening.
* Participants with a history of serologically or biopsy confirmed autoimmune disorders are excluded from this study. As an exception, participants with EATL whose celiac disease is well controlled and who will maintain a strict gluten-free diet are eligible.

Participants with prior autoimmune thyroiditis who are now on stable thyroid replacement therapy are also eligible.

* HTLV I/II positive participants with a history of HTLV-associated myelopathy/tropical spastic paraparesis (TSP)
* Participants who have received prior CD25-directed therapy.
* Current or prior anti-cancer treatment prior to the first dose of study drug as defined below:

  * Any cytotoxic therapy, immunotherapy, antitumor vaccines or monoclonal antibodies within 2 weeks before the start of lymphodepleting chemotherapy.
  * High doses of systemic corticosteroids (>20 mg prednisone or equivalent) 5 days before apheresis and/or 5 days before CAR T cell infusion.
  * Participants who have not reached D+100 following auto-SCT or who have any unresolved Auto-SCT related complications (e.g. pneumonitis).
  * Participants who have undergone prior allogeneic stem cell at any time.
* Participants taking any investigational agents for any disease/ condition.
* Seropositive for human immunodeficiency virus (HIV).
* Active bacterial infections or active viral infections (CMV, syphilis)
* Uncontrolled EBV infection Note: EBV positive test is allowed due to frequent association of active EBV with mature T-cell malignancies, which frequently resolve with improved control of the malignancy. EBV positive participants may be treated with rituximab or biosimilar prior to lymphodepleting chemotherapy at investigator s discretion.
* Active hepatitis C infection.

NOTE: Participants seropositive for hepatitis C virus (HCV) infection must have been treated and cured as defined by undetectable HCV viral load.

-Active hepatitis B infection.

NOTE: Participants that are positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) must have a negative hepatitis B virus polymerase chain reaction (HBV PCR) result <100 IU/mL at screening. Those who are HBV PCR positive are excluded. Those hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive with a negative PCR for hepatitis B will be treated with antivirals designed to prevent hepatitis B reactivation (e.g., entecavir) and have monitoring for hepatitis B reactivation with PCR.

* Participants with current cardiac atrial or cardiac ventricular lymphoma involvement.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, or other clinically significant cardiac disease within 12 months of enrollment.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computer tomography (CT) scan at screening.

NOTE: History of radiation pneumonitis in the radiation field (fibrosis) is allowed.

* History or presence of non-malignant CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* Deep vein thrombosis or pulmonary embolism requiring ongoing systemic anticoagulation
* History of severe immediate hypersensitivity reaction to tocilizumab or any of the agents used in this study
* Participants with second malignancies in addition to their T-cell malignancy are not eligible if the second malignancy has required treatment (including maintenance therapy) within the past 3 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
* Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2044-06-01 (Estimated); Study Completion 2044-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine safety profile of administering autologous CCR4 CAR T cells | 12 weeks
  The number of participants who experience Adverse Events per CTCAE v5.0, by type, grade and frequency of toxicities from time of lymphodepleting regimen through 12 weeks after the last cell infusion.

SECONDARY OUTCOMES:
To determine the feasibility of manufacturing and delivering the targeted dose level of CCR4 CAR T cells to participants | 1 year
  Feasibility will be defined by the successful manufacturing and expansion of the CCR4 CAR T cells for the first 6 participants to satisfy the targeted dose level and meet the requirements of the COA.
Overall survival (OS) | After confirmed disease progression or initiation of new anti-cancer therapy, survival assessed every 3-6 months (+/- 28 days) up to 15 years.
  OS will be assessed in each group and reported using the Kaplan-Meier method.
Duration of response (DOR) and Progression-free survival (PFS) | weeks 4, 12, then every 3 months until Month 12, then at Months 18 and 24 then every 6 months until Month 60 then yearly, after cell infusion, until progression or up to 15 years post cell infusion.
  DOR and PFS will be assessed with radiographic findings and reported using the Kaplan-Meier method.
Complete response rate (CR), Partial response rate (PR) and Overall response rate (ORR=CR+PR) | Weeks 4, 12, then every 3 months until Month 12, then at Months 18 and 24 after cell infusion.
  CR, PR and ORR will be assessed with radiographic findings and reported using the Kaplan-Meier method.
Determine long-term safety profile of autologous CCR4 CAR T cells | Day 0 (cell infusion) up to 15 year after cell infusion
  The long term safety will be assessed by the presence of RCL as well as clinical assessments. RCL samples at 3, 6 and 12 month post- cell infusion then yearly if needed. Once 3 consecutive samples are negative, RCL samples no longer need to be collected. Yearly medical history starting at 12 months to year 15.
Dose Expansion: To determine preliminary efficacy of autologous CCR4 CAR T cells in a limited number of participants at the MTD by assessing the overall response rate (ORR=CR + PR) | Weeks 4, 12, then every 3 months until Month 12 after cell infusion.
  ORR with radiographic findings in each group at baseline, and then best response at weeks 4, 12, then every 3 months until Month 12 after cells.
Dose Escalation: To determine the maximum tolerated dose (MTD) of autologous CCR4 CAR T cells | 28 days from last cell infusion
  The MTD will be determined by the dose found in the 3+3 design to cause design to cause < 33% toxicityas defined by the DLT criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Y Ng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001774-C.html